CLINICAL TRIAL: NCT04644354
Title: The Tocolytic Efficacy of Nifedipine in the Management of Threatened and Advanced Preterm Labor: A Study on 444 Singleton Pregnant Women With Intact Membranes
Brief Title: The Efficacy of Nifedipine in the Management of Preterm Labor
Acronym: BOG/TH/PTL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ethem Unal, M.D., PhD, Associate Prof of Surgery & Surgic (Other Government)
Responsible Party: Sponsor-Investigator, Ethem Unal, M.D., PhD, Associate Prof of Surgery & Surgic, MD, Umraniye Education and Research Hospital
Organization: Umraniye Education and Research Hospital (Other Government)
Other Study IDs: BakirkoyDogumeviTez/2005
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Preterm Labor; Preterm Birth; Preterm Labor Without Delivery; Preterm Labor With Preterm Delivery in Third Trimester; Calcium-Channel Blockers Toxicity; Side Effect of Drug
Keywords: Nifedipine; Tocolytics
MeSH Terms: conditions — Obstetric Labor, Premature; Premature Birth | interventions — Nifedipine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A - Advanced Preterm Labor (aPL): Singleton pregnant women with spontaneous preterm labor at their 23-36 weeks: regular contractions 4 or more in 20 minutes and cervical dilatation at 2 cm and above
  Interventions: Drug: Nifedipine 10 mg
- Group B - Threatened Preterm Labor (tPL): Singleton pregnant women with spontaneous preterm labor at their 23-36 weeks: regular contractions less then 4 in 20 minutes and cervical dilatation less then 2 cm
  Interventions: Drug: Nifedipine 10 mg

INTERVENTIONS:
Drug: Nifedipine 10 mg — For both groups, when preterm labor is diagnosed, 10 mg capsule will be given sublinguially and if it is not effective in 1 hour, the same dose will be repeated again, and the same regimen will be repeated every day till preterm labor ends or proceed to a preterm birth.

SUMMARY:
Preterm labor is one of the problems of obstetrics, and is one of the leading cause of neonatal morbidity and mortality. The incidence of preterm birth is around 7 to 9 %. The preterm baby is prone to respiratory, renal, neurologic and gastrointestinal problems. The correct diagnosis should be followed by the early administration of the most effective tocolytic agent with least side effects for both mother and fetus. Nifedipine, a calcium channel blocker, has gained a world-wide popularity recently since it has the least side-effects on both mother and fetus. In the present study, we aimed to evaluate the success rate of tocolytic agent 'nifedipine' on the spontaneous preterm labor of singeton pregnant women with intact amnionic membrane.

DETAILED DESCRIPTION:
Preterm birth is the main reason of perinatal morbidity and mortality. The main management method of this important problem is to prolong the pregnancy period and to use corticosteroids to prevent fetal pulmonary distress. The most widely studied tocolytic agents, ritodrin, salbutamol and terbutaline are all betamimetics, and they are shown to prolong birth labor till 7 days and do not have any effct on the fetal mortality. However, their maternal side-effects are inevitable and can be mortal. They cause tachycardia, hypotension and some biochemical disturbances. Furthermore, maternal death is possible due to pulmonary edema. These adrenergic agonists are the first line tocolytics, but calcium canal blockers are becoming more popular since they have less side effects and comparable efficacy.

Calcium canal blockers are nonspecific smooth muscle relaxants used in adult hypertension treatment. Their tocolytic effect depends on their inhibition of calcium ions into the myometrial cells. In vitro studies have shown that they have strong relaxant effects on human myometrium. In the present study, our aim is to investigate the effects of nifedipine in our clinic in a period between 2002 and 2005, when it was first used in our clinic as the sıngle tocolytic agent. Its success in preventing preterm labor and its complications in our earlier practice will be noted and this retrospective study will guide us in its current usage, dosages and side-effects.

ELIGIBILITY:
Inclusion Criteria:

* ingleton pregnant women with spontaneous preterm labor at their 23-37 weeks.

Exclusion Criteria:

* Normal pregnant women
* Pregnent women before 23 weeks of gestation
* Pregant women between 23 and 37 weeks of gestation, but with preterm early membrane rupture, chorioamnionitis, preterm labor without cervical change, multiple pregnancy, hypertension, intrauterine growth retardation, fetal anomaly, oligoanhidramniosis, placenta previa, decolman placentaand intrauterine fetal death

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Only singleton pregnent women with preterm labor. All are between 23 and 37 weeks of gestation with intact membranes.
Study Population: Only pregnant women (23-37 weeks) with preterm labor
Sampling Method: Non-Probability Sample
Enrollment: 444 (Estimated)
Dates: Start 2020-12-15 (Estimated); Primary Completion 2020-12-20 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Delay Delivery for 1 day | 1 day
  After start of tocolytic nifedipine, the delay recorded till delivery is only 24 hours
Delay Delivery for 2 days | 2 days
  After start of tocolytic nifedipine, the delay recorded till delivery is 48 hours
Delay Delivery for 3 days | 3 days
  After start of tocolytic nifedipine, the delay recorded till delivery is 72 hours
Delay Delivery for 7 days | 7 days
  After start of tocolytic nifedipine, the delay recorded till delivery is 168 hours
Birth before 34 weeks | till 34 weeks of gestation
  After start of tocolytic nifedipine, the preterm birth occurs before 34 weeks
Birth before 37 weeks | till 37 weeks of gestation
  After start of tocolytic nifedipine, the preterm birth occurs before 37 weeks
Birth after 37weeks | after 37 weeks of gestation-normal birth
  After start of tocolytic nifedipine, the preterm birth occurs after 37 weeks (Normal birth)

CONTACTS AND LOCATIONS:
Overall Officials: Aysun Firat, M.D., Specialist of Obstetrics&Gynecology, Dir, Principal Investigator — Study Director

IPD SHARING:
Plan to Share IPD: Yes
All data will be available at Excel file and be shared by email upon any request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available on December 2020 and will be shared to the end of 2021.
Access Criteria: Anyone who wants to see the data.

REFERENCES:
- [Background] Flenady V, Wojcieszek AM, Papatsonis DN, Stock OM, Murray L, Jardine LA, Carbonne B. Calcium channel blockers for inhibiting preterm labour and birth. Cochrane Database Syst Rev. 2014 Jun 5;2014(6):CD002255. doi: 10.1002/14651858.CD002255.pub2. PMID 24901312
- [Background] de Heus R, Mulder EJ, Visser GH. Management of preterm labor: atosiban or nifedipine? Int J Womens Health. 2010 Aug 9;2:137-42. doi: 10.2147/ijwh.s7219. PMID 21072306
- [Background] Smith GN. What are the realistic expectations of tocolytics? BJOG. 2003 Apr;110 Suppl 20:103-6. doi: 10.1016/s1470-0328(03)00053-3. PMID 12763123
- See also: Principal sponsor ID — https://scholar.google.com.tr/citations?user=6bFlCZwAAAAJ&hl=tr